CLINICAL TRIAL: NCT02220166
Title: Phase II Study on Safety of 60 Days Administration of Triticum Monococcum in Patients With Celiac Disease on Remission in Gluten Free Diet
Brief Title: Safety of Prolonged Administration of Triticum Monococcum in Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Alberto Lanzini, MD PhD, Associate Professor of Gastroenterology, Università degli Studi di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GE-GA2-2010
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Gluten; Gluten free diet; Triticum monococcum
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triticum monococcum (Experimental): 60 days of daily administration of 100 grams of water biscuits of Triticum monococcum
  Interventions: Dietary Supplement: Triticum monococcum

INTERVENTIONS:
Dietary Supplement: Triticum monococcum

SUMMARY:
Preliminary studies on safety profile of Triticum Monococcum (Tm, a variety of Ancient Wheat) have provided conflicting results with some in vitro and ex vivo studies consistent with non toxicity and other suggestive of toxicity. We recently reported results of a single administration of 2.5 grams of Tm in 12 Celiacs in remission on Gluten Free Diet (GFD), while assessing symptoms and changes of intestinal permeability. Although results of intestinal permeability were inconclusive Tm, but not other type of gluten, was clinically well tolerated.

The aim of the present study was to assess safety of 60 days of administration of Tm (100 grams of water biscuits per day accounting for about 6 grams of gluten from Tm) as judged on clinical, serological and histological parameters in Celiac Disease patients on remission after 1 year of GFD.

ELIGIBILITY:
Inclusion Criteria:

* Adult Celiac patients on Gluten Free Diet (GFD) for at least one year
* Strict adherence to GFD
* Negative Celiac related serology
* Normal duodenal Histology defined as Marsh Class 0-II
* Willing to participate and adhere to study protocol
* Sign of the informed consent

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Histologic: 4 duodenal biopsies obtained and classified according to Marsh | Baseline, Day 60
  After 60 days of daily administration of Tm endoscopic biopsies were performed and reviewed by the same experienced pathologist

SECONDARY OUTCOMES:
Clinical: Change in Gastrointestinal Symptom Rating Scale (GSRS) | Baseline, Day 30, Day 60

OTHER OUTCOMES:
Serological: test for immunoglobulin A anti tissue transglutaminases and anti-endomysial | Baseline, Day 30, Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Lanzini, MD, PhD, Study Chair — Università degli Studi di Brescia; Barbara Zanini, MD, PhD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- AO Spedali Civili of Brescia, Brescia, Italy

REFERENCES:
- [Background] Zanini B, Petroboni B, Not T, Di Toro N, Villanacci V, Lanzarotto F, Pogna N, Ricci C, Lanzini A. Search for atoxic cereals: a single blind, cross-over study on the safety of a single dose of Triticum monococcum, in patients with celiac disease. BMC Gastroenterol. 2013 May 24;13:92. doi: 10.1186/1471-230X-13-92. PMID 23706063